CLINICAL TRIAL: NCT00581048
Title: Oxidant Stress and Allergic Asthma
Brief Title: Study on the Role of Treatment With Vitamin E on Asthmatic Responses in Allergic Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryszard T. Dworski, MD, PhD, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#051158; 5K23HL080030-02 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Allergic Asthma
Keywords: Asthma; Allergy; Atopy; Vitamin E; GSTP1; Oxidative stress
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Natural source d-α-tocopheryl acetate (Experimental): 1500 units daily for 16 weeks
  Interventions: Drug: Natural source d-α-tocopheryl acetate

INTERVENTIONS:
Drug: Natural source d-α-tocopheryl acetate — 1500 units daily for 16 weeks
  Other Names: Vitamin E

SUMMARY:
Asthma is a common respiratory disease of unknown etiology which currently affects approximately 7.5 % of the adult population ( ). Asthma is an inflammatory disorder of the airways. Airway inflammation is evident not only in patients with fatal asthma but also in mild asthmatics ( ). Oxidant stress, defined as inadequately controlled generation of toxic reactive oxygen species (ROS) in the cells or tissues is a common feature of inflammation, and has also been documented in asthma ( , ). However, the current understanding of the relationship between the inflammation and the oxidant stress in asthmatic airways is poor. Does oxidant stress contribute to the expression of asthmatic phenotypes independently of inflammation? If so, could asthmatics benefit from supplementation of antioxidants? These questions have been nagging us since our laboratory provided credible evidence of oxidant injury in the airways of allergic asthmatics ( ). The purpose of our study is to more precisely determine 1/ the pathophysiologic role of oxidative stress, and 2/ usefulness of antioxidant therapy using vitamin E in allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Normal health status except for allergic asthma
* Physician diagnosis of mild allergic asthma
* Positive allergen skin tests to common aeroallergens

Exclusion Criteria:

* Use of systemic or high doses of inhaled corticosteroids, >840 mcg of inhaled beclomethasone of its equivalent (as defined in the consensus report (6))
* Past history of severe asthma (as defined in the consensus report (6))
* History of asthma exacerbation within the past month
* History of recent upper respiratory infection within the past month
* Active immunotherapy for allergic diseases
* Significant disease other than allergic asthma and allergic rhinitis, such as coronary disease, hypertension, renal failure, anemia, immunodeficiency, cancer, diabetes
* Present or remote tobacco smoking
* Use of Over The Counter drugs including acetaminophen and pseudoephedrine, herbs, or vitamins
* Psychiatric illness that would make adherence to protocol difficult
* Inability to give informed consent
* Nursing or pregnant women
* Woman planning to become pregnant during the study or not using adequate birth control methods (barrier or hormonal methods)
* H/o sensitivity to tocopherol-derivatives or medications used during bronchoscopy
* Inability to comply with the research protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-12; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Dworski, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Dep. of Medicine, Div. of Allergy, Pulmonary and Critical Care Medicine, Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natural Source d-α-tocopheryl Acetate
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Natural Source d-α-tocopheryl Acetate
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Effect of Natural-source d-α-tocopheryl Acetate on the Baseline and Allergen-induced Levels of F2-isoprostanes in the Bronchoalveolar Lavage Fluid (BAL)
Time Frame: At baseline to after 16-18 weeks of treatment with vitamin E daily
Population: Underlying data was lost. Go to https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3476459 Figure 1 for diagram of results
Arm/Group | Before Treatment, Baseline | After Treatment
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Effect of Treatment With Vitamin E on Airway Reactivity to Methacholine
Time Frame: At baseline and After 16-18 weeks of treatment with vitamin E
Population: Underlying data was lost. Go to https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3476459 Figure 2 for diagram of results
Arm/Group | Before Treatment, Baseline | After Treatment
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Allergen-provoked Concentrations of Th1 and Th2 Cytokines in BAL
Time Frame: baseline to after 16-18 weeks of treatment with vitamin E daily
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Before Treatment, Baseline | After Treatment
Number analyzed (Participants) | 33 | 33
pg/mL
  IL-1B | 0.97 [0.3 to 1.69] | 1.21 [0.52 to 1.98]
  IL-2 | 0.48 [0.2 to 0.99] | 0.69 [0.23 to 1.48]
  IL-3 | 1.6 [0 to 7.7] | 1.4 [0 to 4.5]
  IL-4 | 0.17 [0.03 to 0.57] | 0.045 [0 to 0.2]
  IL-5 | 1.0 [0.33 to 2.9] | 0.8 [0.41 to 13.6]
  IL-6 | 21.5 [5.55 to 111.9] | 17 [4.35 to 94.6]
  IL-9 | 0 [0 to 6.25] | 0 [0 to 5.6]
  IL-10 | 0.53 [0.29 to 1.09] | 0.7 [0.25 to 1.18]
  IL-12 | 0.05 [0.002 to 0.21] | 0.165 [0.078 to 0.41]
  IL-13 | 0.6 [0.4 to 1.96] | 1.0 [0.075 to 3.6]
  TNF-a | 2.76 [0.65 to 11.6] | 3.02 [0.96 to 14.3]
  INF-Y | 0.49 [0.23 to 0.96] | 0.7 [0.3 to 1.65]
  CXCL8 | 44.0 [25.2 to 93.5] | 53.2 [31.0 to 92.3]
  CCL5 | 3.0 [1.36 to 7.11] | 2.3 [1.71 to 8.34]
  CCL11 | 1.0 [0 to 4.02] | 2.70 [0 to 5.45]

4. Secondary Outcome: Allergen-provoked Concentrations of Immunoglobulin E (IgE) in BAL
Time Frame: baseline to after 16-18 weeks of treatment with vitamin E daily
Measure: Median (Inter-Quartile Range); unit: UI/ml
Arm/Group | Before Treatment, Baseline | After Treatment
Number analyzed (Participants) | 33 | 33
UI/ml | 4.05 [2.81 to 10.8] | 3.65 [2.87 to 12.9]

ADVERSE EVENTS:
Arm/Group | Natural Source d-α-tocopheryl Acetate
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes